CLINICAL TRIAL: NCT04316507
Title: Oncologist-Initiated Cancer Genetic Testing for Pancreatic Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 437-2019
Record Dates: First submitted 2020-03-10; First posted 2020-03-20 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncologist led genetic counselling and testing (Experimental): All subjects receive Oncologist Led Genetic Counselling and Testing
  Interventions: Procedure: Genetic Counselling and Testing

INTERVENTIONS:
Procedure: Genetic Counselling and Testing — Oncologist-initiated brief genetic counselling and testing

SUMMARY:
Pancreatic cancer (PC) has a dismal prognosis. Approximately 10% of PC patients carry a germline pathogenic variant in a cancer susceptibility gene, whose identification can lead to better treatments for the patient and participation in cancer prevention programs for their family members. Conventional genetic testing for PC patients is based on the family history of cancer, and may take up to six months from the point of meeting with the treating physician to receiving the results from a genetic counsellor. The median overall survival for these patients is 6 - 12 months, which may prevent them from having the genetic testing in the first place, or from receiving further targeted treatments. Patients with PC need a more comprehensive knowledge of their disease for better treatment planning. This includes genetic testing in absence of family history of cancer.

The investigators designed a one year study to assess the feasibility of medical oncologist initiated cancer genetic testing for all newly diagnosed PC patients unselected by family history.

For patients with negative genetic testing, no further testing will be ordered after the disclosure of results. Patients with positive genetic testing results will be informed and referred to Cancer Genetics Clinic. The investigators expect to enroll 100 patients in 1 year. Patients will be asked to complete satisfaction questionnaires according to the Satisfaction with Genetic Counseling Scale in multiple time points (pre-testing, post-testing, at 6 months and at 12 months). Designated oncologists will be asked to evaluate the process using the Oncologist Satisfaction Survey after every five counseled patients.

Three primary objectives will include 1) assessment of the turnaround time for genetic testing results; 2) assessment of patient satisfaction; 3) assessment of oncologist's satisfaction. Secondary objectives will include assessment of association between genetic testing results and types of treatment and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* • Newly diagnosed exocrine pancreatic cancer

  * Patient consents to blood draw and genetic testing
  * Treating oncologist at Odette Cancer Centre
  * No conditions that would prevent patients from completing the study-related questionnaires or understanding the consent process
  * Valid phone number
  * Email address to send link to online family history questionnaire
  * Treating physician agrees to complete the referrals

Exclusion Criteria:

* Patient declines genetic testing
* Blood transfusion within the past month
* Allogenic bone marrow transplantation
* History of comprehensive panel genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Days from decision to test to receiving genetic test results | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No